CLINICAL TRIAL: NCT03152786
Title: Evaluating the Effect of ADRB2 Blockers on PKA/BAD/CREB Signaling in Patients Undergoing Prostatectomy
Brief Title: Propranolol Hydrochloride in Treating Patients With Prostate Cancer Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PIs not interested in continuing with the trial.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00043227; NCI-2017-00788 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 85716 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-12

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Propranolol; propranolol CR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (propranolol hydrochloride) (Experimental): Patients receive propranolol hydrochloride PO 2 hours prior to standard of care prostatectomy.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Propranolol Hydrochloride; Other: Questionnaire Administration; Other: Survey Administration
- Group II (no treatment) (Active Comparator): Patients receive no treatment prior to standard of care prostatectomy.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Propranolol Hydrochloride — Given PO
  Other Names: Inderal; Innopran XL
  Arms: Group I (propranolol hydrochloride)
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies how well propranolol hydrochloride works in treating patients with prostate cancer who are undergoing surgery. When stressed, the body makes a molecule that may prevent tumor cells from dying, and propranolol hydrochloride may affect the signals in cells that cause tumor cells survival and death.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare activation of ADRB2/PKA/BAD signaling pathway in the prostate glands of men two hours after taking or not taking propranolol hydrochloride (propranolol) prior to prostatectomy, as indicated by phosphorylated CREB.

SECONDARY OBJECTIVES:

I. To compare activation of ADRB2/PKA/BAD signaling pathway in the prostate glands of men two hours after taking or not taking propranolol prior to prostatectomy as indicated by phosphorylated BAD.

II. To determine the difference in candidate transcript levels associated with ADRB2/PKA activation between individuals two hours after taking propranolol or not taking propranolol prior to prostatectomy.

III. To determine plasma propranolol levels in individuals taking propranolol two hours after administration prior to prostatectomy.

IV. To determine if plasma catecholamine levels in men with prostate cancer can be used as a biomarker to identify patients who show activation of ADRB2 signaling pathway in prostate tumors.

V. To determine perceived stress level differences in men with prostate cancer prior to surgery to examine possible association between perceived stress level and catecholamine levels in blood and activation of ADRB2 pathway in tumors.

VI. To determine perceived distress level differences in men with prostate cancer prior to surgery to examine possible association between distress level and catecholamine levels in blood and activation of ADRB2 pathway tumors.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients receive propranolol hydrochloride orally (PO) 2 hours prior to standard of care prostatectomy.

GROUP II: Patients receive no treatment prior to standard of care prostatectomy.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer undergoing prostatectomy
* Individuals able to understand and willing to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Men taking propranolol on a daily for any reason are excluded
* Men with baseline systolic blood pressure (SBP) < 110 or heart rate (HR) < 60
* Men unable to swallow pills
* History of current or past medical or psychiatric illness that would make participation difficult or not feasible at the discretion of the principal investigator or co-investigators

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Hemal, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 15, 2019 to June 8, 2021
Period: Overall Study
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
Started | 23 | 23
Completed | 21 | 22
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment) | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.35 (6.21) | 64.61 (64.61) | 66.48 (6.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 23 | 23 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Mean Level of CREB Phosphorylation
Description: Determined using western blot in prostate tissue from men. CREB is a type of protein that binds to DNA in very specific places. CREB is related to long-term memory formation in the brain and is important in the formation of spatial memory. Phosphorylation alters the structural conformation of a protein, causing it to become activated, deactivated, or otherwise modifying its function. The level of CREB phosphorylation is an indicator of BAD activity.
Time Frame: 2 hours after taking or not taking propranolol prior to prostatectomy
Population: levels of total CREB signal were below detection limit in missing participants
Measure: Mean (Standard Deviation); unit: West blot band intensity,arbitrary units
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
Number analyzed (Participants) | 6 | 5
West blot band intensity,arbitrary units | 1.34 (.33) | 1.43 (.46)

2. Secondary Outcome: BAD Phosphorylation
Description: Will be assessed by western blot in prostate tissue from men. BAD is a protein that plays a critical role in cell survival. Phosphorylation alters the structural conformation of a protein, causing it to become activated, deactivated, or otherwise modifying its function. This analysis shows how much phosphorylation of BAD protein is happening in cells.
Time Frame: 2 hours after taking or not taking propranolol prior to prostatectomy
Population: BAD phosphorylation not detected
Measure: Mean (Standard Deviation); unit: kDa
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
Number analyzed (Participants) | 21 | 22
kDa | 0 (0) | 0 (0)

3. Secondary Outcome: Distress Score - National Comprehensive Cancer Network Distress Thermometer Questionnaire
Description: Will be measured by The Distress Thermometer from men.
  The NCCN Distress Thermometer (DT) is a one-item, 11-point Likert scale represented on a visual graphic of a thermometer that ranges from 0 (no distress) to 10 (extreme distress), with which patients indicate their level of distress over the course of the week prior to assessment. Scoring scale ranges from 0 (no distress) to 10 (extreme distress) with higher scores indicating more distress.
Time Frame: On the day of surgery before taking propranolol, prior to prostatectomy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
Number analyzed (Participants) | 20 | 23
score on a scale | 3.6 (2.3) | 2.7 (2.6)

4. Secondary Outcome: Levels of Transcripts That Reflect ADRB2/PKA Activation
Description: Difference in levels of transcripts that reflect ADRB2/PKA activation will be measured by real-time polymerase chain reaction in prostate tissue from men.
Time Frame: 2 hours after taking or not taking propranolol prior to prostatectomy
Population: insufficient material for RNA extraction
Measure: Mean (Standard Deviation); unit: relative gene expression
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
Number analyzed (Participants) | 21 | 22
relative gene expression | NA (NA) — insufficient material for RNA extraction | NA (NA) — insufficient material for RNA extraction

5. Secondary Outcome: Plasma Catecholamine Levels (Including Epinephrine)
Description: Will be measured by enzyme-linked immunosorbent assay from men. 2-sample t-tests will be calculated to compare the groups who were randomized to receive propranolol (yes/no). Descriptive statistics will be calculated for each measure within each group. These statistics include n, mean, standard deviations and 95% confidence intervals.
Time Frame: 2 hours after taking or not taking propranolol prior to prostatectomy
Population: one blood sample was missing during Epi measurement
Measure: Mean (Standard Deviation); unit: nano mole (nm) per liter (L)
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
Number analyzed (Participants) | 7 | 8
nano mole (nm) per liter (L) | 0.36 (0.22) | 0.34 (0.22)

6. Secondary Outcome: Plasma Propranolol Levels
Description: Will be measured by fluorometric detection from men. 2-sample t-tests will be calculated to compare the groups who were randomized to receive propranolol (yes/no). Descriptive statistics will be calculated for each measure within each group. These statistics include n, mean, standard deviations and 95% confidence intervals.
Time Frame: 2 hours after taking or not taking propranolol prior to prostatectomy
Population: Number of samples collected for analysis.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
Number analyzed (Participants) | 8 | 8
nanograms per milliliter (ng/ml) | 10.89 (4.58) | 0.00 (0.00)

7. Secondary Outcome: Self-perceived Stress
Description: Will be measured by The Perceived Stress Questionnaire from men. The perceived stress questionnaire is a set of 4 questions asking participants about their feelings/problems with stress over the last two weeks. Scoring scale ranges from 0 to 16 with higher scores indicating a higher level of stress.
Time Frame: On the day of surgery before taking propranolol, prior to prostatectomy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
Number analyzed (Participants) | 20 | 23
score on a scale | 7.4 (2.3) | 8.2 (1.4)

ADVERSE EVENTS:
Time Frame: from baseline up to about 2 hours
Arm/Group | Group I (Propranolol Hydrochloride) | Group II (no Treatment)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT03152786/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03152786/ICF_000.pdf